CLINICAL TRIAL: NCT02748616
Title: A Clinical Trial for the Off Label Use of Ursodiol for the Prevention of Recurrent C. Difficile Colitis and Diarrhea
Brief Title: C. Difficile and Ursodiol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-01348
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Diarrhea
Keywords: Colitis; Bile
MeSH Terms: conditions — Diarrhea; Colitis | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ursodiol (Experimental): Subjects will begin to take 300 mg Ursodiol following Visit #1 and continue for a total of 8 (eight) weeks.
  Interventions: Drug: Ursodiol

INTERVENTIONS:
Drug: Ursodiol — Subjects will begin to take 300 mg Ursodiol 2 (two) weeks after Visit #1 for a total of 8 (eight) weeks.
  Other Names: Urso

SUMMARY:
In vitro findings have established that ursodeoxycholic acid is a surrogate for deoxycholic acid in preventing the growth of C. difficile, and interrupting recurrence. Investigators will administer ursodeoxycholic acid for two months, beginning with Metronidazole and/or Vancomycin (8 to 10 days), antibiotics currently used for the treatment of acute C.Difficile infection. Ursodeoxycholic acid prevents c.difficile recurrence by (a) directly suppressing the growth of C. Difficile and (b) permitting restoration of normal fecal bile acid composition (80% deoxycholic acid) to maintain growth suppression.

DETAILED DESCRIPTION:
The non-investigational reference therapies, Metronidazole, Vancomycin and fidaxomicin , are FDA-approved antibiotics currently in use today because of their effectiveness in suppressing the growth of C. difficile and therefore quickly eliminating the colitis and diarrhea. However, they do not promote the restoration of the normal bacterial flora. Therefore, when medication is stopped, the C. difficile colitis returns. In vitro findings have established that ursodeoxycholic acid is a surrogate for deoxycholic acid in preventing the growth of C. difficile, and interrupting recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with recurrent C. difficile colitis
* 18 years of age and older
* Capable of giving informed consent

Exclusion Criteria:

* Patients with other gastrointestinal problems prone to cause diarrhea if they cannot be controlled for the period of the study. Lactose intolerance or gluten enteropathy are not an exclusion provide that the potential subject is asymptomatic and can be expected to adhere to the appropriate dietary regimen.
* Patients with contraindications to metronidazole or vancomycin and/or ursodiol tablets or components of the formulations.
* Patients not available for long-term follow-up (2 months) by their physician will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Javitt, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ursodiol
Started | 9
Completed | 2
Not Completed | 7
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2
Not completed — Did Not Complete Ursodial Course | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ursodiol
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 52 [28 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With Return Toward a Normal Fecal Bile Acid Pattern
Time Frame: 2 months
Measure: Number; unit: percentage of participants
Arm/Group | Ursodiol
Number analyzed (Participants) | 2
percentage of participants | 100

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Ursodiol
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT02748616/Prot_SAP_000.pdf